CLINICAL TRIAL: NCT03305081
Title: Patient Compliance With Long-Acting Reversible Contraception Administration Immediately and Early Postpartum Versus Interval Postpartum
Brief Title: Patient Compliance With Long-Acting Reversible Contraception Administration
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRBNet ID 628424-1
Record Dates: First submitted 2014-11-24; First posted 2017-10-09 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate or early placement (Experimental): Immediate or early placement of levonorgestrel IUD, copper IUD, or etonorgestrel sub dermal implant (within 48 hours) postpartum
  Interventions: Device: Levonorgestrel IUD, copper IUD, etonorgestrel implant
- Interval placement (Active Comparator): Interval (4-6 weeks) postpartum placement of levonorgestrel IUD, copper IUD, or etonorgestrel sub dermal implant
  Interventions: Device: Levonorgestrel IUD, copper IUD, etonorgestrel implant

INTERVENTIONS:
Device: Levonorgestrel IUD, copper IUD, etonorgestrel implant — Long-acting reversible contraception

SUMMARY:
This a randomized control trial to identify if patients who desire LARC are more likely to have success receiving the desired form of contraception if it is placed a) during the postpartum hospital stay, either in the immediate or early postpartum period, versus b) during the interval postpartum period as previously done.

DETAILED DESCRIPTION:
Randomized control trial with control group receiving LARC at 6 weeks postpartum and the study group receiving LARC in the immediate or early postpartum period. Outcomes will be measured by those who receive or do not receive LARC either in the hospital after delivery versus 6 weeks postpartum in accordance with the study subjects' randomized designation. Secondary outcomes of bleeding profile and satisfaction will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, desires LARC postpartum

Exclusion Criteria:

* Medical contraindication to desired LARC, vaginal delivery complicated by fourth degree perineal laceration, history of pelvic inflammatory disease, uterine infection

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2015-12-21 (Actual); Study Completion 2016-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Junya, MD, Principal Investigator — Tulane University School of Medicine
Locations (1):
- Tulane Department of Obstetrics and Gynecology, New Orleans, Louisiana, United States

REFERENCES:
- [Result] Brito MB, Ferriani RA, Quintana SM, Yazlle ME, Silva de Sa MF, Vieira CS. Safety of the etonogestrel-releasing implant during the immediate postpartum period: a pilot study. Contraception. 2009 Dec;80(6):519-26. doi: 10.1016/j.contraception.2009.05.124. Epub 2009 Jul 10. PMID 19913145
- [Result] Celen S, Sucak A, Yildiz Y, Danisman N. Immediate postplacental insertion of an intrauterine contraceptive device during cesarean section. Contraception. 2011 Sep;84(3):240-3. doi: 10.1016/j.contraception.2011.01.006. Epub 2011 Feb 21. PMID 21843687
- [Result] Chen BA, Reeves MF, Hayes JL, Hohmann HL, Perriera LK, Creinin MD. Postplacental or delayed insertion of the levonorgestrel intrauterine device after vaginal delivery: a randomized controlled trial. Obstet Gynecol. 2010 Nov;116(5):1079-87. doi: 10.1097/AOG.0b013e3181f73fac. PMID 20966692
- [Result] Dahlke JD, Terpstra ER, Ramseyer AM, Busch JM, Rieg T, Magann EF. Postpartum insertion of levonorgestrel--intrauterine system at three time periods: a prospective randomized pilot study. Contraception. 2011 Sep;84(3):244-8. doi: 10.1016/j.contraception.2011.01.007. Epub 2011 Feb 24. PMID 21843688
- [Result] Grimes DA, Lopez LM, Schulz KF, Van Vliet HA, Stanwood NL. Immediate post-partum insertion of intrauterine devices. Cochrane Database Syst Rev. 2010 May 12;(5):CD003036. doi: 10.1002/14651858.CD003036.pub2. PMID 20464722
- [Result] Guazzelli CA, de Queiroz FT, Barbieri M, Torloni MR, de Araujo FF. Etonogestrel implant in postpartum adolescents: bleeding pattern, efficacy and discontinuation rate. Contraception. 2010 Sep;82(3):256-9. doi: 10.1016/j.contraception.2010.02.010. Epub 2010 Mar 29. PMID 20705154
- [Result] Levi E, Cantillo E, Ades V, Banks E, Murthy A. Immediate postplacental IUD insertion at cesarean delivery: a prospective cohort study. Contraception. 2012 Aug;86(2):102-5. doi: 10.1016/j.contraception.2011.11.019. Epub 2012 Jan 20. PMID 22264666
- [Result] Shukla M, Qureshi S; Chandrawati. Post-placental intrauterine device insertion--a five year experience at a tertiary care centre in north India. Indian J Med Res. 2012 Sep;136(3):432-5. PMID 23041736
- [Result] Stuart GS, Bryant AG, O'Neill E, Doherty IA. Feasibility of postpartum placement of the levonorgestrel intrauterine system more than 6 h after vaginal birth. Contraception. 2012 Apr;85(4):359-62. doi: 10.1016/j.contraception.2011.08.005. Epub 2011 Sep 28. PMID 22067759

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate or Early Placement | Interval Placement
Started | 25 | 20
Completed | 15 | 5
Not Completed | 10 | 15
Not completed — Lost to Follow-up | 10 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate or Early Placement | Interval Placement | Total
Number analyzed (Participants) | 25 | 20 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 23 | 19 | 42
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 20 | 45
Patients Presenting to the Office or Hospital [Count of Participants; unit: Participants] | 25 | 20 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Women With Placement of LARC
Description: The outcome will be measured by the number of participants with LARC placement. The total number of women who expressed a desire to have postpartum contraception placed and randomized to the appropriate arm will be assessed.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate or Early Placement | Interval Placement
Number analyzed (Participants) | 25 | 20
Participants | 10 | 2

2. Secondary Outcome: Patient Satisfaction With Method of LARC Using LARC Survey
Description: Number of patients satisfied with LARC obtained by LARC survey at 6-weeks, 12-weeks postpartum, and 6 months postpartum. Patients identify Yes/No response via telephone survey asking, "Are you satisfied with this form of contraception?". Satisfaction determined if subject answers "Yes". A single value was calculated at the end of the study by summation at all three time points.
Time Frame: 6 Weeks, 12 weeks postpartum, 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate or Early Placement | Interval Placement
Number analyzed (Participants) | 25 | 15
Participants | 10 | 2

ADVERSE EVENTS:
Arm/Group | Immediate or Early Placement | Interval Placement
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/20
Other Adverse Events (participants affected / at risk) | 0/25 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes